CLINICAL TRIAL: NCT06135272
Title: Evaluation of Three Different Minimally Invasive Techniques for Management of Enamel Opacities in Patients With Molar Incisor Hypomineralization "Randomized Controlled Clinical Trial"
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Collaborators: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Hagar Mahmoud Mohie, PhD researcher, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PED23-4D
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Molar Incisor Hypomineralization
Keywords: MIH; Molar Incisor Hypomineralization; enamel opacities; giomer varnish; ICON; Resin infiltration; Clinpro xt; resin modified glass ionomer varnish
MeSH Terms: conditions — Molar Hypomineralization; enamel opacities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Resin infiltration
  Interventions: Drug: Resin infiltration
- Group B (Experimental): Resin modified glass ionomer varnish
  Interventions: Drug: Resin modified glass ionomer varnish
- Group C (Experimental): Light cured giomer varnish
  Interventions: Drug: Light cured giomer varnish

INTERVENTIONS:
Drug: Resin infiltration — Icon Resin Infiltration as minimally invasive technique
  Arms: Group A
Drug: Resin modified glass ionomer varnish — Resin modified glass ionomer varnish as minimally invasive technique
  Arms: Group B
Drug: Light cured giomer varnish — Light cured giomer varnish as minimally invasive technique
  Arms: Group C

SUMMARY:
The controlled clinical trial will be done to evaluate Resin infiltration, Resin modified glass ionomer varnish and Light cured giomer varnish as minimally invasive techniques for management of enamel opacities of patients with molar incisor hypomineralization. Variation in mineral density of the enamel opacity , ,Hypersensitivity, Color change of the enamel opacity, Quality of life of the patient, Parent Satisfaction will be evaluated preoperatively and at 1, 3,6,12 and 18 months of follow up.

DETAILED DESCRIPTION:
A total of 75 patients will be selected according to the eligibility criteria from the Pediatric Dentistry and Dental Public Health outpatient clinic, Faculty of Dentistry, Ain Shams University.

A Full detailed medical and dental history will be obtained from the parent and a clinical examination will be performed using a dental mirror and a dental explorer under LED illumination and after dryness of the teeth to make sure that the patients fulfill the inclusion criteria.

After explaining the aim of the study, benefits, possible risks and rights to the patients and their parents. A signed informed consent of the parents as well as child's assent, outlined by the Ethical Committee, Faculty of Dentistry, Ain Shams University will be obtained prior to the conduction of the study. • The patients will be randomly equally allocated into three treatment groups (25 patients/ group): Group (A): patients will receive resin infiltration. Group (B): patients will receive resin modified glass ionomer varnish. Group (C): patients will receive a light cured giomer varnish.

Pre-operative procedures:

* Patients will be interviewed the oral health related quality of life questionnaire and it will be assessed prior treatment.
* Mineral density of the tooth will be measured using laser fluorescence.
* Teeth will be tested for sensitivity using recent validated test.
* Tooth color will be measured using vita easy shade.

Clinical procedures

- All teeth will be cleaned using prophylaxis paste and brush.

Group A:

1. Local anesthesia administration and rubber dam isolation.
2. Application of 15% hydrochloric acid gel (Icon etch) on affected enamel for two minutes and it will be washed for 30 seconds.
3. Application of 99% ethanol (Icon dry) for 30 seconds then it will be dried using air-water tip.
4. Application of Icon resin on the affected enamel surface and it will be left for three minutes to allow penetration.
5. The resin will be light cured for 40 seconds then the excess will be removed.
6. The Icon resin will be reapplied for one minute then light cured for 40 seconds.
7. The tooth will be polished using composite polishing discs.

Group B:

1. Application of 37% phosphoric acid gel on affected enamel for 15 seconds then rinse and dry for five seconds.
2. The material will be dispensed and mixed for 15 seconds.
3. The material will be applied to the affected tooth surface and light cured for 20 seconds.
4. The excess will be removed using a moist cotton.

Group C:

1. One drop of the active of the material will be mixed with one container of the base using a disposable brush.
2. A thin layer of the mixture will be applied on the affected enamel surface after drying and it will be left undistributed for three seconds
3. The material will be light cured for 10 seconds.

   * The patients will be counselled to follow a proper diet and instructed about oral hygiene measures using soft tooth brush and fluoridated tooth paste twice daily.
   * All patients will be scheduled to receive dental treatment for other dental findings at the Department of Pediatric Dentistry, Faculty of Dentistry, Ain Shams University.

The patient will be followed at 1, 3,6,12 and 18 months for evaluation of:

1. Mineral density of the opacity
2. Hypersensitivity
3. Color change of the opacity
4. Quality of life of the patient
5. Parent Satisfaction

Statistical Analysis All data will be tabulated, summarized and statistically analyzed using software SPSS (Statistical Packages for Social Sciences).

ELIGIBILITY:
Inclusion Criteria:

* Patient with molar incisor hypomineralization having at least one incisor and/or molar mildly affected.
* Patient's age ranges from 6 to 10 years old.
* The affected tooth has demarcated opacity without post eruptive enamel breakdown.
* No cavitated lesion is related to the defect or previous restorative or preventive treatment.
* The tooth is free from any symptoms of irreversible pulp inflammation.

Exclusion Criteria:

* Children who are physically or mentally disabled or having any medical condition that will affect or complicate the treatment.
* Incisors previously subjected to trauma that might lead to loss of tooth structure or compromised the pulp vitality.
* Loss of tooth structure due to caries.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Variation in mineral density | It will be evaluated preoperatively and at 1, 3,6,12 and 18 months follow up.
  Variation in mineral density of the enamel opacity using laser fluorescence.
Hypersensitivity | It will be evaluated pre operative and at 1, 3,6,12 and 18 months follow up.
  Hypersensitivity using VAS scale

SECONDARY OUTCOMES:
Color change of the enamel opacity | It will be evaluated preoperatively and at 1, 3,6,12 and 18 months of follow up.
  Color change of the enamel opacity using Vita easy shade
Quality of life of the patient | It will be evaluated preoperatively and at 1, 3,6,12 and 18 months of follow up.
  Quality of life of the patient using Child Perceptions Questionnaire (CPQ)
Parent Satisfaction | It will be evaluated preoperatively and at 1, 3,6,12 and 18 months of follow up.
  Parent Satisfaction using Parental-Caregivers Perceptions Questionnaire (P- CPQ )

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No